CLINICAL TRIAL: NCT00097357
Title: A Phase 2 Randomized, Double-Blinded (BMS-562247 and Enoxaparin), Active-Controlled (Enoxaparin and Warfarin), Parallel-Arm, Dose-Response Study of the Oral Factor Xa Inhibitor BMS-562247 in Subjects Undergoing Elective Total Knee Replacement Surgery
Brief Title: BMS-562247 in Subjects Undergoing Elective Total Knee Replacement Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-010
Record Dates: First submitted 2004-11-22; First posted 2004-11-23 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-11

CONDITIONS: Venous Thrombosis; Pulmonary Embolism
Keywords: Prevention of deep vein thrombosis and pulmonary embolism; Preventive therapy
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — apixaban; Enoxaparin; Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- A1 (Experimental): Apixaban: 2.5 mg, BID
  PLUS
  Enoxaparin Placebo
  Interventions: Drug: Apixaban; Drug: Enoxaparin Placebo
- A2 (Experimental): Apixaban: 5 mg, BID
  PLUS
  Enoxaparin Placebo
  Interventions: Drug: Apixaban; Drug: Enoxaparin Placebo
- A3 (Experimental): Apixaban: 10 mg, BID
  PLUS
  Enoxaparin Placebo
  Interventions: Drug: Apixaban; Drug: Enoxaparin Placebo
- A4 (Experimental): Apixaban: 5 mg, QD
  PLUS
  Enoxaparin Placebo
  Interventions: Drug: Apixaban; Drug: Enoxaparin Placebo
- A5 (Experimental): Apixaban: 10 mg, QD
  PLUS
  Enoxaparin Placebo
  Interventions: Drug: Apixaban; Drug: Enoxaparin Placebo
- A6 (Experimental): Apixaban: 20 mg, QD
  PLUS
  Enoxaparin Placebo
  Interventions: Drug: Apixaban; Drug: Enoxaparin Placebo
- E1 (Active Comparator): Enoxaparin: 30 mg
  PLUS
  Apixaban Placebo
  Interventions: Drug: Enoxaparin; Drug: Apixaban Placebo
- W1 (Active Comparator): Warfarin: 5 mg tablets dose titrated to a targeted INR of 1.8 to 3.0
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — Tablets, Oral, 12 +/- 2 days
  Other Names: BMS-562247
  Arms: A1; A2; A3; A4; A5; A6
Drug: Enoxaparin — Injection, SQ, Q12H, 12 +/- 2 days
  Arms: E1
Drug: Warfarin — Tablets, Oral, QD, 12 +/- 2 days
  Arms: W1
Drug: Enoxaparin Placebo — Injection, SQ, BID, 12 +/- 2 days
  Arms: A1; A2; A3; A4; A5; A6
Drug: Apixaban Placebo — Tablets, Oral, BID, 12 +/- 2 days
  Arms: E1

SUMMARY:
The purpose of this study is to learn if BMS-562247 can prevent blood clots in the legs and lungs in men and women following unilateral total knee replacement surgery. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective unilateral total knee replacement surgery.
* Willing and able to undergo bilateral ascending contrast venography.
* Able to inject (by self or caregiver) study medication subcutaneously.

Exclusion Criteria:

* Women of childbearing potential.
* Women who are pregnant or breastfeeding.
* Under some conditions, subjects weighing more than 300 lbs. (136kg) and/or Body Mass Index (BMI) >=35 kg/m2

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1238 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Determine the dose-response relationship among the 3 QD and 3 BID doses of BMS-562247 on the composite endpoint of adjudicated VTE events and all-cause death in subjects treated with study medication for 12 +/-2 days following surgery | throughout the study

SECONDARY OUTCOMES:
Assess the effect of QD and BID dose of BMS-562247 vs subcutaneous 30 mg q12h enoxaparin and warfarin on the composite endpoint of adjudication VTE events and all-cause death in subjects treated for 12 +/-2 days following surgery | throughout the study
Assess the effect of each QD and BID dose of BMS-562247 versus subcutaneous 30 mg q12h enoxaparin and oral warfarin on the incidence of adjudicated major bleeding events in subjects treated with study medication for 12 +/-2 days following surgery | throughout the study
Assess the effect of each QD and BID dose of BMS-562247 versus subcutaneous 30 mg q12h enoxaparin and oral warfarin on the incidence of adjudicated minor bleeding events in subjects treated with study medication for 12 +/-2 days following surgery | throughout the study
To determine the pharmacokinetic (PK) profile of BMS-562247 and the relationship to dose and dose schedule | throughout the study

CONTACTS AND LOCATIONS:
Locations (147):
- United States (72):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Northport, Alabama
  - Local Institution, Phoenix, Arizona
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Beverly Hills, California
  - Local Institution, Encinitas, California
  - Local Institution, Fountain Valley, California
  - Local Institution, La Jolla, California
  - Local Institution, La Mesa, California
  - Local Institution, Long Beach, California
  - Local Institution, Montclair, California
  - Local Institution, Oakland, California
  - Local Institution, Pasadena, California
  - Local Institution, Sacramento, California
  - Local Institution, San Bernardino, California
  - Local Institution, San Diego, California
  - Local Institution, Santa Monica, California
  - Local Institution, Torrance, California
  - Local Institution, Wildomar, California
  - Local Institution, Yuba City, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Hartford, Connecticut
  - Local Institution, Bay Pines, Florida
  - Local Institution, Brandon, Florida
  - Local Institution, Clearwater, Florida
  - Local Institution, DeLand, Florida
  - Local Institution, Fort Myers, Florida
  - Local Institution, Hollywood, Florida
  - Local Institution, Melbourne, Florida
  - Local Institution, Pensacola, Florida
  - Local Institution, Sarasota, Florida
  - Local Institution, St. Petersburg, Florida
  - Local Institution, Tallahassee, Florida
  - Local Institution, Winter Park, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Cumming, Georgia
  - Local Institution, Decatur, Georgia
  - Local Institution, Suwanee, Georgia
  - Local Institution, Boise, Idaho
  - Local Institution, Meridian, Idaho
  - Local Institution, Galesburg, Illinois
  - Local Institution, Springfield, Illinois
  - Local Institution, Wichita, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Madisonville, Kentucky
  - Local Institution, Covington, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Newton, Massachusetts
  - Local Institution, Port Huron, Michigan
  - Local Institution, Jackson, Mississippi
  - Local Institution, Buffalo, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Monroe, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Youngstown, Ohio
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Havertown, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Lubbock, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Newport News, Virginia
  - Local Institution, Seattle, Washington
  - Local Institution, Marshfield, Wisconsin
- Argentina (5):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital fEDERAL, Buenos Aires
  - Local Institution, Prov. Buenos Aires, Buenos Aires
  - Local Institution, Godoy Cruz, Mendoza Province
  - Local Institution, Mendoza, Mendoza Province
- Australia (10):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Chermside, Queensland
  - Local Institution, Gold Coast, Queensland
  - Local Institution, Herston, Queensland
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Clayton, Victoria
  - Local Institution, East Ringwood, Victoria
  - Local Institution, Geelong, Victoria
  - Local Institution, Windsor, Victoria
- Canada (23):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Red Deer, Alberta
  - Local Institution, Kelowna, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Dartmouth, Nova Scotia
  - Local Institution, Ajax, Ontario
  - Local Institution, Burlington, Ontario
  - Local Institution, Greater Sudbury, Ontario
  - Local Institution, Newmarket, Ontario
  - Local Institution, Niagara Falls, Ontario
  - Local Institution, Oakville, Ontario
  - Local Institution, Richmond Hill, Ontario
  - Local Institution, St. Catharines, Ontario
  - Local Institution, Thunder Bay, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Welland, Ontario
  - Local Institution, Weston, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Ste-foy, Quebec
  - Local Institution, Victoriaville, Quebec
- Denmark (5):
  - Local Institution, Frederiksberg
  - Local Institution, Herlev
  - Local Institution, Hørsholm
  - Local Institution, Silkeborg
  - Local Institution, Slagelse
- Israel (8):
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Kfar Saba
  - Local Institution, Petah Tikva
  - Local Institution, Ramat Gan
  - Local Institution, Rehovot
  - Local Institution, Tel Aviv
  - Local Institution, Ẕerifin
- Mexico (13):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Tijuana, Baja California Sur
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Hermosillo, Sonora
  - Local Institution, México, State of Mexico
  - Local Institution, Tampico, Tamps, Tamaulipas
  - Local Institution, Jalapa, Veracruz
  - Local Institution, Veracruz, Veracruz
  - Local Institution, Mérida, Yucatán
- Poland (10):
  - Local Institution, Bialystock
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Piekary Śląskie
  - Local Institution, Radom
  - Local Institution, Sosnowiec
  - Local Institution, Szczecin
  - Local Institution, Szczecin Zdunowo
  - Local Institution, Warsaw
- Local Institution, Ponce, Puerto Rico